CLINICAL TRIAL: NCT04424316
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLINDED, PLACEBO-CONTROLLED TRIAL TO EVALUATE THE EFFICACY AND SAFETY OF A RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE IN INFANTS BORN TO WOMEN VACCINATED DURING PREGNANCY
Brief Title: A Trial to Evaluate the Efficacy and Safety of RSVpreF in Infants Born to Women Vaccinated During Pregnancy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671008; 2019-002943-85 (EudraCT Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory Tract infection; RSV; Vaccine; Maternal
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSVpreF vaccine (Experimental): RSVpreF
  Interventions: Biological: RSVpreF
- Placebo dose (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSVpreF — RSV vaccine (RSVpreF)
  Arms: RSVpreF vaccine
Biological: Placebo — Placebo
  Arms: Placebo dose

SUMMARY:
This randomized, double-blinded, placebo-controlled Phase 3 study is designed to evaluate the efficacy and safety of maternal immunization with RSVpreF against medically attended lower respiratory tract illness (MA-LRTI) in infants.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blinded, placebo-controlled study to assess the efficacy, safety, and immunogenicity of RSVpreF or placebo (1:1 randomization) in infants born to healthy women vaccinated during pregnancy, as well as the safety and immunogenicity in the pregnant women. This will be a global study which will span multiple RSV seasons.

ELIGIBILITY:
Inclusion Criteria - Maternal Participants:

* Healthy women ≤49 years of age who are between 24 0/7 and 36 0/7 weeks of gestation on the day of planned vaccination, with an uncomplicated, singleton pregnancy, who are at no known increased risk for complications.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Receiving prenatal standard of care based on country requirements.
* Had a fetal anomaly ultrasound examination performed at ≥18 weeks of pregnancy with no significant fetal abnormalities observed.
* Determined by medical history, physical examination, and clinical judgment to be appropriate for inclusion in the study.
* Documented negative HIV antibody test, syphilis test, and hepatitis B virus (HBV) surface antigen test during this pregnancy and prior to randomization (Visit 1).
* Intention to deliver at a hospital or birthing facility where study procedures can be obtained.
* Expected to be available for the duration of the study and can be contacted by telephone during study participation.
* Participant is willing to give informed consent for her infant to participate in the study.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol OR If the maternal participant is illiterate, a thumbprinted informed consent must be obtained, which must be signed and dated by an impartial witness who was present throughout the entire informed consent process confirming that the maternal participant has been informed of all pertinent aspects of the study.

Inclusion Criteria -Infant Participants:

* Evidence of a signed and dated ICD signed by the parent(s)/legal guardian(s) OR If the infant participant's maternal participant/parent(s)/legal guardian(s) is illiterate, a thumbprinted informed consent must have been obtained, which must have been signed and dated by an impartial witness who was present throughout the entire informed consent process confirming that the maternal participant/parent(s)/legal guardian(s) has been informed of all pertinent aspects of the study for herself (maternal participant) and her fetus/infant prior to taking part in the study.
* Parent(s)/legal guardian(s) willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria - Maternal Participants:

* Prepregnancy body mass index (BMI) of >40 kg/m2. If prepregnancy BMI is not available, the BMI at the time of the first obstetric visit during the current pregnancy may be used.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product or any related vaccine.
* Current pregnancy resulting from in vitro fertilization.
* Current pregnancy complications or abnormalities at the time of consent that will increase the risk associated with the participation in and completion of the study, including but not limited to the following:

  * Preeclampsia, eclampsia, or uncontrolled gestational hypertension.
  * Placental abnormality.
  * Polyhydramnios or oligohydramnios.
  * Significant bleeding or blood clotting disorder.
  * Endocrine disorders, including untreated hyperthyroidism or untreated hypothyroidism. This also includes disorders of glucose intolerance (eg, diabetes mellitus type 1 or 2) antedating pregnancy or occurring during pregnancy if uncontrolled at the time of consent.
  * Any signs of premature labor with the current pregnancy or having ongoing intervention (medical/surgical) in the current pregnancy to prevent preterm birth.
* Prior pregnancy complications or abnormalities at the time of consent, based on the investigator's judgment, that will increase the risk associated with the participation in and completion of the study, including but not limited to the following:

  * Prior preterm delivery ≤34 weeks' gestation.
  * Prior stillbirth or neonatal death.
  * Previous infant with a known genetic disorder or significant congenital anomaly.
* Major illness of the maternal participant or conditions of the fetus that, in the investigator's judgment, will substantially increase the risk associated with the maternal or infant participant's participation in, and completion of, the study or could preclude the evaluation of the maternal participant's response (includes positive serologic testing for regional endemic conditions assessed during routine maternal care, as per local standards of care and obstetric recommendations).
* Congenital or acquired immunodeficiency disorder, or rheumatologic disorder or other illness requiring chronic treatment with known immunosuppressant medications, including monoclonal antibodies, within the year prior to enrollment.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participation in other studies involving investigational drug(s) within 28 days prior to consent and/or during study participation.
* Receipt of monoclonal antibodies within the year prior to enrollment or the use of systemic corticosteroids for >14 days within 28 days prior to study enrollment. Permitted treatments include the receipt of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) monoclonal antibodies, prednisone doses of <20 mg/day for ≤14 days and, inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids.
* Current alcohol abuse or illicit drug use. Note: Marijuana use is not considered an exclusion criterion for the study when elicited in participant screening, though it may be considered illicit in some locales.
* Receipt of blood or plasma products or immunoglobulin (Ig), from 60 days before investigational product administration, or planned receipt through delivery, with 1 exception, Rho(D) immune globulin (eg, RhoGAM), which can be given at any time.
* Previous vaccination with any licensed or investigational RSV vaccine or planned. Note: Licensed COVID-19 vaccines or COVID-19 vaccines authorized for temporary or emergency use will not be prohibited during the course of this study.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.
* Participants who are breastfeeding at the time of enrollment.

Exclusion Criteria -Infant Participants:

o Infant who is a direct descendant (eg, child or grandchild) of the study personnel.

Ages: 0 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Healthy women ≤49 years of age who are between 24 and 36 weeks of gestation on the day of planned vaccination, with an uncomplicated, singleton pregnancy, who are at no known increased risk for complications.
Enrollment: 14727 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (459):
- United States (359):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Endocrinology and Internal Medicine Associates, PC, Birmingham, Alabama
  - OB/GYN Associates of Alabama, PC, Birmingham, Alabama
  - Sharp and Stone OB/GYN PC, Birmingham, Alabama
  - St Vincent's Hospital, Birmingham, Alabama
  - Children's of Alabama, Birmingham, Alabama
  - UAB Women & Infants Center - UAB Medicine, Birmingham, Alabama
  - University of Alabama at Birmingham/Center for Women's Reproductive Health, Birmingham, Alabama
  - Cullman Clinical Research, Inc, Cullman, Alabama
  - Cullman Primary Care, PC, Cullman, Alabama
  - Cullman Regional, Cullman, Alabama
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Springhill Medical Center, Mobile, Alabama
  - Velocity Clinical Research, Gulfport, Mobile, Alabama
  - Velocity Clinical Research - Pheonix, Phoenix, Arizona
  - Valleywise Comprehensive Health Center Women's Clinic, Phoenix, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - Mesquite Pediatrics, Tucson, Arizona
  - Watching Over Mothers and Babies, Tucson, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Banner University Medical Center ( North Campus ), Tucson, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - St. Bernards OBGYN Associates, Jonesboro, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - The Children's Clinic of Jonesboro, PA, Jonesboro, Arkansas
  - Century Research Institute, Bellflower, California
  - Chowchilla Medical Center, Chowchilla, California
  - Loma Linda University Pediatric Clinic - Highland, Highland, California
  - Century Research Institute, Huntington Park, California
  - Matrix Clinical Research, Huntington Park, California
  - Chemidox Clinical Trials, Lancaster, California
  - Leonard S. Kurian, M.D., A Medical Corporation, Lancaster, California
  - Women & Infants Pavilion, Antelope Valley Hospital, Lancaster, California
  - Loma Linda University Adventist Health Sciences Center, Loma Linda, California
  - Loma Linda University Faculty Medical Clinics, Loma Linda, California
  - Loma Linda University Pediatric Clinics, Loma Linda, California
  - Loma Linda Unversity Children's Hospital, Loma Linda, California
  - Long Beach Clinical Trials, Long Beach, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - St Mary Medical Center, Long Beach, California
  - Century Research Institute, Los Angeles, California
  - Matrix Clinical Research.., Los Angeles, California
  - East LA Doctors Hospital, Los Angeles, California
  - Hollywood Presbyterian Medical Center, Los Angeles, California
  - White Memorial Medical Center, Los Angeles, California
  - Peter Morton Medical Building, Los Angeles, California
  - Ronald Reagan UCLA Medical Center Drug Information Center Dept, Los Angeles, California
  - Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Affiliated Physician Practice, Madera, California
  - Charles E. Ugwu-Oju, M.D., F.A.C.O.G., Obstetrics & Gynecology, Madera, California
  - Madera Community Hospital, Madera, California
  - Madera Family Medical Group, Madera, California
  - Monterey Park Hospital, Monterey Park, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Stanford University, Palo Alto, California
  - Fomat- Raymond Poliakin, MD., Thousand Oaks, California
  - Carey Chronis, MD, Ventura, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Anschutz Inpatient Pavilion 2, Aurora, Colorado
  - University of Colorado AO1, Aurora, Colorado
  - University of Colorado Hospital Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital Outpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - University of Colorado Leprino Building, Aurora, Colorado
  - University of Colorado Research II Building, Aurora, Colorado
  - Delta Memorial Hospital, Delta, Colorado
  - Colorado Canyon's Hospital, Fruita, Colorado
  - Boeson Research, Grand Junction, Colorado
  - Dino-Peds, Grand Junction, Colorado
  - Women's Health Care of Western Colorado, Grand Junction, Colorado
  - Community Hospital, Grand Junction, Colorado
  - SCL St. Mary's Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Yale School Medicine Church Street Research Unit, New Haven, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - North Shore Medical Center, Miami, Florida
  - Citadelle Clinical Research, North Miami Beach, Florida
  - A1 Imaging of Aventura, North Miami Beach, Florida
  - Baldwin Pediatrics, Panama City, Florida
  - Emerald Coast Obstetrics and Gynecology, Panama City, Florida
  - Emerald Coast Pediatrics, Panama City, Florida
  - Gulf Coast Regional Medical Center, Panama City, Florida
  - Rainbow Pediatrics, Panama City, Florida
  - Rainbow Pediatrics, Panama City Beach, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Investigational Drug Service, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Piedmont Columbus Regional Midtown, Columbus, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - 1st Choice Urgent Care & Family Medicine, Blackfoot, Idaho
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Grove Creek Medical Center, Blackfoot, Idaho
  - ASR, LLC, Boise, Idaho
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Luke's Boise Medical Center, Boise, Idaho
  - West Valley Medical Center, Caldwell, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Mountain View Hospital, Idaho Falls, Idaho
  - The Pediatric Center, Idaho Falls, Idaho
  - Saltzer Health, Meridian, Idaho
  - St. Luke's Meridian Medical Center, Meridian, Idaho
  - Saltzer Health, Nampa, Idaho
  - ASR, LLC, Nampa, Idaho
  - St. Alphonsus Medical Center- Nampa, Nampa, Idaho
  - St. Luke's Nampa Medical Center, Nampa, Idaho
  - Pocatello Women's Health Clinic, Pocatello, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - 1st Choice Urgent Care, Pocatello, Idaho
  - Clinical Research Prime Rexburg, Rexburg, Idaho
  - Elite Clinical Trials LLLP, Rexburg, Idaho
  - Madison Memorial Hospital, Rexburg, Idaho
  - The Pediatric Center, Rigby, Idaho
  - Dupont Pediatrics, Fort Wayne, Indiana
  - Women's Health Advantage, Fort Wayne, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - Mcfarland Clinic PC, Ames, Iowa
  - McFarland Clinic, P.C., Ames, Iowa
  - The Iowa Clinic, Ankeny, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - The Iowa Clinic, P.C., West Des Moines, Iowa
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Owensboro Health Regional Hospital, Owensboro, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - The Women's Pavillion, P.S.C, Owensboro, Kentucky
  - Alexandria Cardiology Clinic - Secondary Research Site, Alexandria, Louisiana
  - Cambridge Medical Trials - Main Research Site, Alexandria, Louisiana
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Rabie Clinic for Women, Alexandria, Louisiana
  - Rapides Regional Medical Center Labor and Delivery, Alexandria, Louisiana
  - Lakeview Regional Medical Center, Covington, Louisiana
  - St. Tammany Parish Hospital, Covington, Louisiana
  - Velocity Clinical Research, Covington, Louisiana
  - Ochsner Health Center - West Bank, Gretna, Louisiana
  - North Oaks Medical Center, Hammond, Louisiana
  - North Oaks Obstetrics & Gynecology, Hammond, Louisiana
  - North Oaks Rural Health Clinic, Hammond, Louisiana
  - MedPharmics LLC, Lafayette, Louisiana
  - Crescent City Physicians and Obstetrics, Metairie, Louisiana
  - MedPharmics LLC, Metairie, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ochsner Health Center for Children, New Orleans, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Slidell Memorial Hospital, Slidell, Louisiana
  - Velocity Clinical Research, Slidell, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Investigational Pharmacy Service, Boston, Massachusetts
  - C.S. Mott Center, Detroit, Michigan
  - Hutzel-Harper Women's Hospital, Detroit, Michigan
  - University Health Center, Detroit, Michigan
  - Wayne State University Physician Group, Southfield, Michigan
  - Velocity Clinical Research, Gulfport, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Baer Pediatrics, St Louis, Missouri
  - KDB Enterprises, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Boeson Research (BUT), Butte, Montana
  - St James Healthcare, Butte, Montana
  - Benefis Health System, Great Falls, Montana
  - Origin Health GTF, Great Falls, Montana
  - Boeson Research (GTF), Great Falls, Montana
  - Marcus Daly Memorial Hospital, Hamilton, Montana
  - Boeson Research (HLN), Helena, Montana
  - St Peters Health, Helena, Montana
  - Boeson Reseach (KAL), Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - The Birth Center, Missoula, Montana
  - Boeson Research LLC, Missoula, Montana
  - Boeson Research, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Community Physicians Group-Maternal Fetal Medicine, Missoula, Montana
  - St Luke Community Clinic - Ronan, Ronan, Montana
  - North Valley Hospital, Whitefish, Montana
  - Grand Island Regional Medical Center, Grand Island, Nebraska
  - CHI Health St. Francis, Grand Island, Nebraska
  - Meridian Clinical Research, LLC, Grand Island, Nebraska
  - Mary Lanning, Hastings, Nebraska
  - Meridian Clinical Research, Hastings, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Midwest Children's Health Research Institute., Lincoln, Nebraska
  - Bryan Health, Lincoln, Nebraska
  - Midwest Childrens Health Research Institute, Lincoln, Nebraska
  - Women's Health Care Center of Williamsburg, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Jaffe Family Womens Care Center, Camden, New Jersey
  - Pediatrics at Sheridan Pavilion- Three Cooper Plaza, Camden, New Jersey
  - Cooper Faculty OBGYN at Cherry Hill, Cherry Hill, New Jersey
  - Saint Peters University Hospital, New Brunswick, New Jersey
  - Cooper Faculty OBGYN at Sewell, Sewell, New Jersey
  - MedPharmics, Albuquerque, New Mexico
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Velocity Clinical Research, Albuquerque, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - New York Presbyterian of Queens Hospital, Flushing, New York
  - Theresa Lang Children's Ambulatory Center, Flushing, New York
  - Fresh Meadows Family Health Center, Fresh Meadows, New York
  - Hollis Women's Center, Hollis, New York
  - Jackson Heights Family Health Center, Jackson Heights, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Women's Contemporary Care, Mineola, New York
  - Columbia Doctors, New York, New York
  - Audubon Clinic, New York, New York
  - Center for Prenatal Pediatrics, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Herbert Irving Pavilion, New York, New York
  - Morgan Stanley Childrens Hospital, New York, New York
  - Meridian Clinical Research LLC, Vestal, New York
  - UNC OB/GYN at Panther Creek (recruitment, randomization, administration of IP), Cary, North Carolina
  - UNC Children's Hospital (Pediatric follow up), Chapel Hill, North Carolina
  - UNC Healthcare (recruitment, randomization, administration of IP), Chapel Hill, North Carolina
  - UNC OB/GYN at Weaver Crossing (recruitment, randomization, administration of IP), Chapel Hill, North Carolina
  - Duke Children's Primary Care - Roxboro Street, Durham, North Carolina
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University., Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - FirstHealth Clinical Trials, Pinehurst, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Sandhills Pediatrics, Seven Lakes, North Carolina
  - Sandhills Pediatrics, Southern Pines, North Carolina
  - FirstHealth Southern Pines Women's Health Center, Southern Pines, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center Department of Obstetrics and Gynecology, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - HWC Women's Research Center, LLC, Englewood, Ohio
  - UC Health West Chester Hospital, West Chester, Ohio
  - Integris Yukon Hospital, Yukon, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - OBGYN Associates of Erie, Erie, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Reading Hospital - Children's Health Center, West Reading, Pennsylvania
  - Reading Hospital - Women's Health Center, West Reading, Pennsylvania
  - Reading Hospital-Family Health Care Center, West Reading, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Bon Secours St. Francis Hospital, Charleston, South Carolina
  - Charleston 0B/GYN, Charleston, South Carolina
  - Coastal Pediatric Research, Charleston, South Carolina
  - Prisma Health-Upstate Office of Maternal Fetal Medicine, Greenville, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Lowcountry Womens Specialists, Summerville, South Carolina
  - Summerville Medical Center, Summerville, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Sanford Obstetrics and Gynecology Clinic (Recruitment, Consenting, IP Administration, and Follow Up), Sioux Falls, South Dakota
  - Sanford Obstetrics and Gynecology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center (Main Hospital), Sioux Falls, South Dakota
  - Sanford Women's Health Plaza (Recruitment, Consenting, and Follow Up), Sioux Falls, South Dakota
  - Premier Medical Group, Clarksville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Health Arlington Memorial Hospital, Arlington, Texas
  - Ventavia Research Group, LLC, Arlington, Texas
  - Medical City Arlington (Women's Hospital), Arlington, Texas
  - St. David's Medical Center, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Center for Women''s Health and Birthcare, Beaumont, Texas
  - Christus St. Elizabeth Hospital, Beaumont, Texas
  - Gadolin Research, LLC, Beaumont, Texas
  - Texas Health Harris Methodist Hospital Hurst-Euless-Bedford, Bedford, Texas
  - Child Care Pediatrics, P.A., Burleson, Texas
  - Ventavia Research Group LLC, Burleson, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Ventavia Research Group LLC, Dallas, Texas
  - Wise Health System Dectaur, Decatur, Texas
  - Cline Pediatrics, Dickinson, Texas
  - Doctor's Hospital Womens Hospital, Edinburg, Texas
  - South Texas Health System- Edinburg, Edinburg, Texas
  - 8th Avenue Obstetrics & Gynecology, Fort Worth, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Texas Health Harris Methodist Hospital Fort Worth, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Texas Health Harris Methodist Hospital Southwest, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Chisholm Trail Pediatrics, Georgetown, Texas
  - FMC Science, Georgetown, Texas
  - St. David's Georgetown Hospital, Georgetown, Texas
  - Baylor Scott & White of Grapevine (Hospital), Grapevine, Texas
  - Ventavia Research Group, LLC, Grapevine, Texas
  - Hany H. Ahmed, MD, Houston, Texas
  - HG Pediatrics, Houston, Texas
  - Van Tran Family Clinic, Houston, Texas
  - Ventavia Research Group, LLC, Houston, Texas
  - Memorial Hermann Memorial City, Houston, Texas
  - UT Health Women's Research Center at Memorial City, Houston, Texas
  - HCA: The Women's Hospital of Texas, Houston, Texas
  - Javara Inc., Houston, Texas
  - Privia Medical Group Gulf Coast, PLLC, Houston, Texas
  - Texas Center for Drug Development, Inc, Houston, Texas
  - AdventHealth Family Medicine Rural Health Clinic, Inc., Lampasas, Texas
  - FMC Science, Lampasas, Texas
  - Maximos Ob/Gyn, League City, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Diagnostic Clinic of Longview (Hollybrook), Longview, Texas
  - Diagnostic Clinic of Longview (Medical Circle), Longview, Texas
  - Longview Regional Medical Center, Longview, Texas
  - Rio Grande Regional Hospital, McAllen, Texas
  - South Texas Health System- McAllen, McAllen, Texas
  - Dr. Ruben Aleman and Associates, McAllen, Texas
  - Medical City Plano, Plano, Texas
  - Texas Health Presbyterian Hospital Plano, Plano, Texas
  - Ventavia Research Group LLC, Plano, Texas
  - St. Luke's Baptist Hospital, San Antonio, Texas
  - Tekton Research, LLC., San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Medical City Weatherford, Weatherford, Texas
  - Ventavia Research Group, Weatherford, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - Old Farm Obstetrics & Gynecology, LLC, Salt Lake City, Utah
  - Holladay Family Practice, Salt Lake City, Utah
  - St. Marks Hospital, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Sentara Leigh Hospital, Norfolk, Virginia
  - The Group for Women, Norfolk, Virginia
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Clinical Research Partners, LLC, North Chesterfield, Virginia
  - Virginia Commonwealth Univeristy Health Systems-Children's Pavilion, Richmond, Virginia
  - Virginia Commonwealth University Health System-Main Hospital, Richmond, Virginia
  - Virginia Commonwealth University Health System-Nelson Clinic, Richmond, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - VCU Health Adult Outpatient Pavillion, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Tidewater Physicians for Women, Virginia Beach, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - UW Neighborhood Ravenna Clinic, Seattle, Washington
  - UW Neighborhood South Lake Union Clinic, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - UW Midwives Clinic at Northwest Outpatient Medical center, Seattle, Washington
  - University of Washington Medical Center- Montlake, Seattle, Washington
  - UW Neighborhood Shoreline Clinic, Shoreline, Washington
  - MultiCare Health System - Mary Bridge Children's Health Center, Tacoma, Washington
  - Multicare Health System-Multicare Women's Center Tacoma, Tacoma, Washington
  - Multicare Health System-Pediatrics Northwest, Tacoma, Washington
  - Multicare Health System-Tacoma General Hospital, Tacoma, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - Cabell Huntington Hospital, Huntington, West Virginia
  - Marshall Health, Huntington, West Virginia
  - University Physicians and Surgeons dba Marshall Health Department of Obstetrics and Gynecology, Huntington, West Virginia
  - University Physicians and Surgeons dba Marshall Health Department of Pediatrics, Huntington, West Virginia
  - Marshfield Medical Center - Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
- Argentina (8):
  - Clínica del Niño y la Madre, Mar del Plata, Buenos Aires
  - Hospital Italiano de Rosario, Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Instituto de Maternidad y Ginecologia: "Nuestra Senora de las Mercedes", San Miguel de Tucumán, Tucumán Province
  - Sanatorio Mater Dei, Buenos Aires
  - Centro de Investigación Clinica OSECAC, Buenos Aires
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, CABA
  - Hospital Publico Materno Infantil, Salta
- Australia (5):
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Monash Children's Hospital, Clayton, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Telethon Kids Institute, Nedlands, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- Brazil (4):
  - Hospital Universitario/GAMP - Grupo de Apoio a Medicina Preventiva e a Saude Publica, Canoas, Rio Grande do Sul
  - Hospital Moinhos de Vento - HMV, Porto Alegre, Rio Grande do Sul
  - Maternidade Darcy Vargas, Joinville, Santa Catarina
  - Clinica de Alergia Martti Antila S/S Ltda./ CMPC - Consultoria Medica e Pesquisa Clinica, Sorocaba, São Paulo
- Canada (3):
  - Canadian Center for Vaccinology - IWK Health Centre, Halifax, Nova Scotia
  - CHU Sainte-Justine, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
- Chile (10):
  - Hospital Base San José de Osorno (Servicio de Obstetricia y Ginecología), Osorno, Los Lagos Region
  - Centro de Capacitación e Investigaciones Clínicas (CCIC), Santiago, Santiago Metropolitan
  - Clinica Universidad de los Andes, Santiago, Santiago Metropolitan
  - Satellite (Deliveries): Hospital San Juan de Dios (Maternidad), Santiago, Santiago Metropolitan
  - Instituto de Investigaciones Materno Infantil (IDIMI), Santiago, Santiago Metropolitan
  - Deliveries (satellite): Hospital San Jose, Santiago, Santiago Metropolitan
  - Grupo Estudios Clínicos Infectología Respiratoria, Santiago, Santiago Metropolitan
  - Deliveries (satellite): Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Santiago Metropolitan
  - Hospital Padre Hurtado, Santiago, Santiago Metropolitan
- Denmark (4):
  - Aarhus Universitetshospital, Aarhus N
  - Nordsjællands Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Odense Universitets Hospital, Odense
- Finland (8):
  - MeVac, Helsinki
  - Kokkola Vaccine Research Clinic, Kokkola
  - Oulu Vaccine Research Clinic, Oulu
  - Tampereen yliopisto Oulun Rokotetutkimusklinikka, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinajoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- Japan (12):
  - Fukui Aiiku Hospital, Fukui-shi, Fukui
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Kuwana City Medical Center, Kuwana-shi, Mie-ken
  - Sendai City Hospital, Sendai, Miyagi
  - National Hospital Organization Beppu Medical Center, Beppu, Oita Prefecture
  - Social Medical Corporation KARIYUSHIKAI Heartlife Hospital, Nakagami-gun, Okinawa
  - Osaka Habikino Medical Center, Habikino, Osaka
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Saitama City hospital, Saitama
  - Shizuoka General Hospital, Shizuoka
- Mexico (5):
  - Asociacion Mexicana para la Investigacion Clinica, A. C., Pachuca, Hidalgo
  - Arke SMO S.A. de C.V., Cuauhtémoc, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Hospital General de Durango, Durango
  - Arke SMO S.A. de C.V., Veracruz
- Netherlands (3):
  - Spaarne Gasthuis (Kennemer Gasthuis), Hoofddorp
  - Diakonessenhuis Utrecht, Utrecht
  - University Medical Center Utrecht, Utrecht
- New Zealand (9):
  - Botany Downs Primary Birthing Unit, Golflands, Auckland
  - Papakura Primary Birthing Unit, Papakura North, Auckland
  - Middlemore Hospital, Papatoetoe, Auckland
  - Pukekohe Primary Birthing Unit, Pukekohe, Auckland
  - New Zealand Clinical Research (Christchurch), Christchurch, Canterbury
  - Optimal Clinical Trials Ltd, Auckland
  - Aotearoa Clinical Trials Trust (ACTT), Auckland
  - Christchurch Hospital (Canterbury District Health Board), Christchurch
  - Capital, Coast and Hutt Valley District- Wellington Regional Hospital, Wellington
- Asian Hospital and Medical Center, Muntinlupa City, National Capital Region, Philippines
- South Africa (11):
  - JOSHA Research, Bloemfontein, Free State
  - Wits RHI Shandukani Research Centre, Johannesburg, Gauteng
  - Into Research, West Wing Medical Centre, Pretoria, Gauteng
  - Setshaba Research Centre, Soshanguve, Gauteng
  - University of the Witwatersrand Vaccines & Infectious Diseases Analytics (VIDA), Soweto, Gauteng
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - MRC Unit on Child and Adolescent Health, Cape Town, Western Cape
  - Khayelitsha Satellite Site: Michael Mapongwana Community Health Centre, Khayelitsha, Western Cape
  - FAMCRU, University of Stellenbosch, Paediatric, Parow Valley, Western Cape
  - Kraaifontein Satellite site, Cape Town
  - Worcester Satellite site, Worcester
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruna
  - Hospital de Antequera, Antequera, Malaga
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Madrid Puerta del Sur Mostoles, Móstoles
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (5):
  - Hsinchu MacKay Memorial Hospital, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan District
- The Gambia (2):
  - Medical Research Council Unit the Gambia at the London School of Hygiene & Tropical Medicine, Fajara KMC
  - Medical Research Council Unit the Gambia at the London School of Hygiene & Tropical Medicine (LSHTM), Sukuta

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bolanos R, Araos R, Gonzalez C, Sepulveda D, Falconi JF, Averin A, Atwood M, Quinn E, Law AW, Mendes D. Cost-effectiveness of strategies using preventive interventions to protect infants in Chile from respiratory syncytial virus. Expert Rev Vaccines. 2025 Dec;24(1):904-913. doi: 10.1080/14760584.2025.2562201. Epub 2025 Oct 2. PMID 40958705
- [Derived] Ilangovan K, Radley D, Patton M, Shittu E, Lino MM, Goulas C, Swanson KA, Anderson AS, Gurtman A, Munjal I. Integrated Analysis of the Safety Experience in Adults with the Bivalent Respiratory Syncytial Virus Prefusion F Vaccine. Vaccines (Basel). 2025 Aug 1;13(8):827. doi: 10.3390/vaccines13080827. PMID 40872913
- [Derived] Simoes EAF, Pahud BA, Madhi SA, Kampmann B, Shittu E, Radley D, Llapur C, Baker J, Perez Marc G, Barnabas SL, Fausett M, Adam T, Perreras N, Van Houten MA, Kantele A, Huang LM, Bont LJ, Otsuki T, Vargas SL, Gullam J, Tapiero B, Stein RT, Polack FP, Zar HJ, Staerke NB, Padilla MD, Richmond PC, Sarwar UN, Baber J, Koury K, Lino MM, Kalinina EV, Li W, Cooper D, Anderson AS, Swanson KA, Gurtman A, Munjal I; MATISSE (Maternal Immunization Study for Safety and Efficacy) Clinical Trial Group. Efficacy, Safety, and Immunogenicity of the MATISSE (Maternal Immunization Study for Safety and Efficacy) Maternal Respiratory Syncytial Virus Prefusion F Protein Vaccine Trial. Obstet Gynecol. 2025 Feb 1;145(2):157-167. doi: 10.1097/AOG.0000000000005816. Epub 2025 Jan 2. PMID 39746212
- [Derived] Madhi SA, Kampmann B, Simoes EAF, Zachariah P, Pahud BA, Radley D, Sarwar UN, Shittu E, Llapur C, Perez Marc G, Maldonado Y, Kachikis A, Zar HJ, Swanson KA, Lino MM, Anderson AS, Gurtman A, Munjal I. Preterm Birth Frequency and Associated Outcomes From the MATISSE (Maternal Immunization Study for Safety and Efficacy) Maternal Trial of the Bivalent Respiratory Syncytial Virus Prefusion F Protein Vaccine. Obstet Gynecol. 2025 Feb 1;145(2):147-156. doi: 10.1097/AOG.0000000000005817. Epub 2025 Jan 2. PMID 39746206
- [Derived] Nazareno AL, Wood JG, Muscatello DJ, Homaira N, Hogan AB, Newall AT. Estimating the cost-effectiveness of maternal respiratory syncytial virus (RSV) vaccination in Australia: A dynamic and economic modelling analysis. Vaccine. 2025 Feb 6;46:126651. doi: 10.1016/j.vaccine.2024.126651. Epub 2024 Dec 28. PMID 39733477
- [Derived] Otsuki T, Akada S, Anami A, Kosaka K, Munjal I, Baber J, Shoji Y, Aizawa M, Swanson KA, Gurtman A. Efficacy and safety of bivalent RSVpreF maternal vaccination to prevent RSV illness in Japanese infants: Subset analysis from the pivotal randomized phase 3 MATISSE trial. Vaccine. 2024 Sep 17;42(22):126041. doi: 10.1016/j.vaccine.2024.06.009. Epub 2024 Jun 8. PMID 38853036
- [Derived] Kampmann B, Madhi SA, Munjal I, Simoes EAF, Pahud BA, Llapur C, Baker J, Perez Marc G, Radley D, Shittu E, Glanternik J, Snaggs H, Baber J, Zachariah P, Barnabas SL, Fausett M, Adam T, Perreras N, Van Houten MA, Kantele A, Huang LM, Bont LJ, Otsuki T, Vargas SL, Gullam J, Tapiero B, Stein RT, Polack FP, Zar HJ, Staerke NB, Duron Padilla M, Richmond PC, Koury K, Schneider K, Kalinina EV, Cooper D, Jansen KU, Anderson AS, Swanson KA, Gruber WC, Gurtman A; MATISSE Study Group. Bivalent Prefusion F Vaccine in Pregnancy to Prevent RSV Illness in Infants. N Engl J Med. 2023 Apr 20;388(16):1451-1464. doi: 10.1056/NEJMoa2216480. Epub 2023 Apr 5. PMID 37018474
- [Derived] Ginsburg AS, Srikantiah P. Respiratory syncytial virus: promising progress against a leading cause of pneumonia. Lancet Glob Health. 2021 Dec;9(12):e1644-e1645. doi: 10.1016/S2214-109X(21)00455-1. Epub 2021 Nov 11. No abstract available. PMID 34774184
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14727 participants were enrolled (7420 maternal participants and 7307 infant participants) in the study.
Groups:
- Maternal Participants: RSVpreF: Study-eligible pregnant women (maternal participants) were randomized to receive a single dose of 120 micrograms (mcg) respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF), intramuscularly (IM) on Day 1 (day of vaccination). Participants were followed up to 6 months after delivery.
- Maternal Participants: Placebo: Maternal participants were randomized to receive placebo matching to RSVpreF as a single dose on Day 1 (day of vaccination). Participants were followed up to 6 months after delivery.
- Infant Participants: RSVpreF: Infant participants born to maternal participants vaccinated with a single dose of 120 mcg RSVpreF were included. Infant participants were all followed up for 12 months after birth, and for infants born to maternal participants during the first year of the study, they were followed up for 24 months after birth.
- Infant Participants: Placebo: Infant participants born to maternal participants who received placebo (matching RSVpreF without active vaccine) were included. Infant participants were all followed up for 12 months after birth, and for infants born to maternal participants during the first year of the study, they were followed up for 24 months after birth.
Period: Overall Study
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo | Infant Participants: RSVpreF | Infant Participants: Placebo
Started (As product administered.) | 3712 (One maternal participant was randomized to placebo arm but received RSVpreF, hence included here.) | 3708 | 3661 (One infant participant born to maternal participant was randomized to placebo arm but received RSVpreF, hence included here.) | 3646
Safety Population (Maternal safety population included all randomized maternal participants who received investigational product. Infant safety population included all infant participants who were born to vaccinated maternal participants.) | 3698 (Received investigational product.) | 3687 (Received investigational product.) | 3659 (Infant born to maternal participants according to investigational product received.) | 3646 (Infant born to maternal participants according to investigational product received.)
Completed | 3516 | 3509 | 3318 | 3294
Not Completed | 196 | 199 | 343 | 352
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 8 | 14
Not completed — Lost to Follow-up | 93 | 88 | 224 | 211
Not completed — No longer met eligibility criteria | 1 | 0 | 0 | 0
Not completed — Other | 15 | 11 | 34 | 45
Not completed — Physician Decision | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 71 | 77 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 74 | 81
Not completed — Randomized but not vaccinated | 13 | 21 | 0 | 0
Not completed — Mother vaccinated but unblinded during study | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Maternal safety population included all randomized maternal participants who received investigational product. Infant safety population included all infant participants who were born to vaccinated maternal participants.
Groups:
- Maternal Participants: RSVpreF: Study-eligible pregnant women (maternal participants) were randomized to receive a single dose of 120 mcg RSVpreF, IM on Day 1 (day of vaccination). Participants were followed up to 6 months after delivery.
- Total: Total of all reporting groups
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo | Infant Participants: RSVpreF | Infant Participants: Placebo | Total
Number analyzed (Participants) | 3698 | 3687 | 3659 | 3646 | 14690
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 3659 | 3646 | 7323
  Between 18 and 65 years | 3689 | 3678 | 0 | 0 | 7367
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3698 | 3687 | 1794 | 1815 | 10994
  Male | 0 | 0 | 1865 | 1831 | 3696
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1063 | 1086 | 1079 | 1081 | 4309
  Not Hispanic or Latino | 2605 | 2568 | 2529 | 2519 | 10221
  Unknown or Not Reported | 30 | 33 | 51 | 46 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 38 | 37 | 42 | 36 | 153
  Asian | 456 | 464 | 446 | 456 | 1822
  Native Hawaiian or Other Pacific Islander | 9 | 12 | 13 | 11 | 45
  Black or African American | 720 | 725 | 706 | 706 | 2857
  White | 2397 | 2375 | 2340 | 2328 | 9440
  More than one race | 30 | 21 | 65 | 59 | 175
  Unknown or Not Reported | 48 | 53 | 47 | 50 | 198

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infant Participants With Medically Attended Lower Respiratory Tract Illness (MA-LRTI) Cases Due to RSV Occurring Within 90 Days After Birth (Efficacy)
Description: Results are presented as confirmed by endpoint adjudication committee. MA-LRTI case: infant with an MA-RTI visit with age related fast breathing (respiratory rate [RR] more than or equal to [>=] 60 breaths per minute [bpm] for less than [<] 2 months of age [<60 days of age], >=50 bpm for >=2 months to <12 months of age, or >=40 bpm for >=12 months to 24 months of age) or oxygen saturation (SpO2) <95 percent (%) or chest wall indrawing and RSV positive test results by reverse transcription-polymerase chain reaction (RT-PCR) testing of midturbinate nasal swab samples.
Time Frame: Within 90 days after birth
Population: Evaluable efficacy - infant population included all infant participants who were born to the maternal participants who received the investigational product to which they were randomized (RSVpreF or placebo) at least 14 days prior to delivery; did not receive palivizumab or another monoclonal antibody targeting RSV; had no major protocol violations and did not have transfusions of more than 20 milliliter/kilogram (mL/kg) of any blood products at <180 days.
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 0.7 | 1.7
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine Efficacy = 57.6, 95% CI 2-sided [31.3 to 74.6]

2. Primary Outcome: Percentage of Infant Participants With MA-LRTI Cases Due to RSV Occurring Within 120 Days After Birth (Efficacy)
Description: Results are presented as confirmed by endpoint adjudication committee. MA-LRTI case: Infant with an MA-RTI visit with age related fast breathing (RR >=60 bpm for <2 months of age [<60 days of age], >=50 bpm for >=2 months to <12 months of age, or >=40 bpm for >=12 months to 24 months of age) or SpO2 <95% or chest wall indrawing and RSV positive test results by RT-PCR testing of midturbinate nasal swab samples.
Time Frame: Within 120 days after birth
Population: Evaluable efficacy - infant population included all infant participants who were born to the maternal participants who received the investigational product to which they were randomized (RSVpreF or placebo) at least 14 days prior to delivery; did not receive palivizumab or another monoclonal antibody targeting RSV; had no major protocol violations and did not have transfusions of more than 20 mL/kg of any blood products at <180 days.
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 1.1 | 2.5
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 54.5, 95% CI 2-sided [33.2 to 69.5]

3. Primary Outcome: Percentage of Infant Participants With MA-LRTI Cases Due to RSV Occurring Within 150 Days After Birth (Efficacy)
Description: as for outcome 2
Time Frame: Within 150 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 1.5 | 3.1
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 50.0, 95% CI 2-sided [30.3 to 64.5]

4. Primary Outcome: Percentage of Infant Participants With MA-LRTI Cases Due to RSV Occurring Within 180 Days After Birth (Efficacy)
Description: as for outcome 2
Time Frame: Within 180 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 1.9 | 3.7
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 49.2, 95% CI 2-sided [31.4 to 62.8]

5. Primary Outcome: Percentage of Infant Participants With Severe MA-LRTI Cases Due to RSV Occurring Within 90 Days After Birth (Efficacy)
Description: Results are presented as confirmed by endpoint adjudication committee. Severe MA-LRTI cases were a subset of MA-LRTI cases, and all severe MA-LRTI cases included MA-LRTI cases. Severe MA-LRTI case was an RSV positively adjudicated event which met the following defined criteria: an infant with an MA-RTI visit and aged associated fast breathing (RR >=70 bpm for <2 months of age [<60 days of age], >=60 bpm for >=2 months to <12 months of age, or >=50 bpm for >=12 months to 24 months of age) or SpO2 <93% or high-flow nasal cannula or mechanical ventilation (i.e., invasive or non-invasive) or intensive care unit (ICU) admission for more than (>) 4 hours or failure to respond/unconscious.
Time Frame: Within 90 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 0.2 | 1.0
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 82.4, 95% CI 2-sided [57.5 to 93.9]

6. Primary Outcome: Percentage of Infant Participants With Severe MA-LRTI Cases Due to RSV Occurring Within 120 Days After Birth (Efficacy)
Description: Results are presented as confirmed by endpoint adjudication committee. Severe MA-LRTI cases were a subset of MA-LRTI cases, and all severe MA-LRTI cases were included MA-LRTI cases. Severe MA-LRTI case was an RSV positively adjudicated event which met the following defined criteria: an infant with an MA-RTI visit and aged associated fast breathing (RR >=70 bpm for <2 months of age [<60 days of age], >=60 bpm for >=2 months to <12 months of age, or >=50 bpm for >=12 months to 24 months of age) or SpO2 <93% or high-flow nasal cannula or mechanical ventilation (i.e., invasive or non-invasive) or ICU admission for >4 hours or failure to respond/unconscious.
Time Frame: Within 120 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 0.4 | 1.4
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 73.5, 95% CI 2-sided [50.3 to 86.8]

7. Primary Outcome: Percentage of Infant Participants With Severe MA-LRTI Cases Due to RSV Occurring Within 150 Days After Birth (Efficacy)
Description: as for outcome 6
Time Frame: Within 150 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 0.5 | 1.7
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 70.5, 95% CI 2-sided [49.4 to 83.6]

8. Primary Outcome: Percentage of Infant Participants With Severe MA-LRTI Cases Due to RSV Occurring Within 180 Days After Birth (Efficacy)
Description: as for outcome 6
Time Frame: Within 180 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases | 0.6 | 2.0
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Vaccine Efficacy = 70.0, 95% CI 2-sided [50.6 to 82.5]

9. Primary Outcome: Percentage of Infant Participants With Adverse Events of Special Interest (AESI) (Safety)
Description: AESI are a subset of targeted medical events based on review of known pharmacology, toxicology findings, possible class effects, published literature, and signals arising from safety data assessments, and on population under study. AESIs were based on targeted medical events associated with pregnant maternal participants and their infants prior to/during delivery and at birth. For infant participants the following were considered as protocol defined AESIs: Preterm birth (born at <37 weeks gestation); birth weight 1001-2500 grams; developmental delay; positive viral (polymerase chain reaction [PCR] or antigen-based) testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), when not reported during MA-RTI visit, were reported as SARS-CoV-2 test positive. Extremely preterm birth (<28 weeks) and extremely low birth weight (=<1000 grams [g]) were reported as serious AESIs.
Time Frame: From birth to 24 months of age
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3659 | 3646
Percentage of participants | 11.9 [10.8 to 13.0] | 10.3 [9.3 to 11.3]

10. Primary Outcome: Percentage of Infant Participants With Neonatal Deaths (Safety)
Description: Neonatal death was defined as the death of a live-born infant that occurred within a month after birth.
Time Frame: Within 1 Month after birth
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3659 | 3646
Percentage of participants | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.3]

11. Primary Outcome: Percentage of Infant Participants With Congenital Malformations/Anomalies (Safety)
Description: Congenital malformations/ anomalies were defined as structural or functional anomalies that occurred during intrauterine life and could be identified prenatally, at birth or later in life.
Time Frame: At birth
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3659 | 3646
Percentage of participants | 5.6 | 6.7

12. Primary Outcome: Percentage of Infant Participants With Other Neonatal Events (Safety)
Description: Other Neonatal problem included dysmaturity, neonatal illness, hospitalization, drug therapies, and neonatal death.
Time Frame: Within 1 Month after birth
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3659 | 3646
Percentage of participants | 6.2 | 5.5

13. Primary Outcome: Number of Infant Participants According to Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) Score at 1 Minute After Birth (Safety)
Description: APGAR was a fast evaluation technique used to evaluate a newborn baby's overall health. APGAR stands for (A) Appearance (skin coloration), (P) Pulse (heart rate), (G) Grimace (reflex response), (A) Activity (muscle tone) and (R) Respiration (breathing). Each component was given a score of 0, 1, or 2; after summing up scores for each component a total possible score was of 0 (worst condition) to 10 (best condition), where higher scores indicate better health. A score of 7 to 10 was good, 4 to <7 was moderate, and <4 was poor.
Time Frame: 1 minute after birth
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3625 | 3606
Participants
  Score <4 | 49 | 44
  Score 4 to <7 | 135 | 124
  Score 7 to 10 | 3441 | 3438

14. Primary Outcome: Number of Infant Participants According to APGAR Score at 5 Minutes After Birth (Safety)
Description: as for outcome 13
Time Frame: 5 minutes after birth
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3618 | 3602
Participants
  Score <4 | 8 | 5
  Score 4 to <7 | 29 | 27
  Score 7 to 10 | 3581 | 3570

15. Primary Outcome: Number of Infant Participants According to APGAR Score at 10 Minutes After Birth (Safety)
Description: as for outcome 13
Time Frame: 10 minutes after birth
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 999 | 999
Participants
  Score <4 | 0 | 0
  Score 4 to <7 | 6 | 4
  Score 7 to 10 | 993 | 995

16. Primary Outcome: Percentage of Infant Participants With Adverse Events (AEs) From Birth to 1 Month of Age (Safety)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From birth to 1 month of age
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3659 | 3646
Percentage of participants | 38.0 [36.4 to 39.6] | 35.4 [33.9 to 37.0]

17. Primary Outcome: Percentage of Infant Participants With Serious Adverse Events (SAEs) and Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Birth Through 6 Months of Age (Safety)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect or that was considered an important medical event. An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From birth to 6 months of age
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3568 | 3558
Percentage of participants
  SAE | 16.7 [15.5 to 17.9] | 16.4 [15.2 to 17.7]
  NDCMC | 1.3 [0.9 to 1.7] | 1.6 [1.2 to 2.1]

18. Primary Outcome: Percentage of Infant Participants With SAEs and NDCMCs From Birth Through 12 Months of Age (Safety)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life threatening required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect or that was considered an important medical event. An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From birth to 12 months of age
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3568 | 3558
Percentage of participants
  SAE | 17.3 [16.1 to 18.6] | 17.2 [15.9 to 18.5]
  NDCMC | 2.1 [1.7 to 2.6] | 2.3 [1.9 to 2.9]

19. Primary Outcome: Percentage of Infant Participants With SAEs and NDCMCs From Birth Through 24 Months of Age (Safety)
Description: as for outcome 18
Time Frame: From birth to 24 months of age
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3659 | 3646
Percentage of participants
  SAE | 19.0 [17.8 to 20.4] | 18.9 [17.6 to 20.2]
  NDCMC | 3.9 [3.3 to 4.6] | 4.5 [3.8 to 5.2]

20. Primary Outcome: Percentage of Maternal Participants With Prespecified Local Reactions Within 7 Days After Vaccination (Safety)
Description: Local reactions included redness, swelling, and pain at injection site and were recorded in electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit= 0.5 centimetre (cm). Redness and swelling were graded as mild (>2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and grade 4 (necrosis or exfoliative dermatitis for redness and necrosis for swelling). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and grade 4 (emergency room visit or hospitalization for the severe pain at the injection site). Grade 4 reactions were classified by the investigator or medically qualified person.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Maternal safety population included all randomized maternal participants who received investigational product. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo
Number analyzed (Participants) | 3678 | 3651
Percentage of participants
  Redness: Any | 7.2 [6.4 to 8.1] | 0.2 [0.1 to 0.4]
  Redness: Mild | 5.0 [4.3 to 5.7] | 0.1 [0.0 to 0.3]
  Redness: Moderate | 2.1 [1.7 to 2.6] | 0.1 [0.0 to 0.3]
  Redness: Severe | 0.1 [0.0 to 0.3] | 0 [0.0 to 0.1]
  Redness: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Swelling: Any | 6.2 [5.4 to 7.0] | 0.2 [0.1 to 0.4]
  Swelling: Mild | 4.1 [3.5 to 4.8] | 0.1 [0.0 to 0.3]
  Swelling: Moderate | 2.0 [1.6 to 2.5] | 0.1 [0.0 to 0.2]
  Swelling: Severe | 0.1 [0.0 to 0.2] | 0 [0.0 to 0.1]
  Swelling: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Pain at injection site: Any | 40.7 [39.1 to 42.3] | 10.2 [9.2 to 11.2]
  Pain at injection site: Mild | 36.1 [34.6 to 37.7] | 9.3 [8.4 to 10.3]
  Pain at injection site: Moderate | 4.5 [3.8 to 5.2] | 0.9 [0.6 to 1.2]
  Pain at injection site: Severe | 0.1 [0.0 to 0.3] | 0 [0.0 to 0.1]
  Pain at injection site: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]

21. Primary Outcome: Percentage of Maternal Participants With Prespecified Systemic Events Within 7 Days After Vaccination (Safety)
Description: Systemic events included: fever, fatigue, headache, nausea, muscle pain, joint pain, vomiting and diarrhea and were recorded by participants in an e-diary. Fever was defined as an oral temperature >=38.0 degree Celsius [C]) and classified as mild (38.0 to 38.4), moderate (38.5 to 38.9), severe (39.0 to 40.0) and grade 4 (>40.0 degree C). Headache, nausea, fatigue, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily activity). Vomiting: mild (1-2 times in 24 hours [H]), moderate (>2 times in 24 H), severe (required intravenous [IV] hydration). Diarrhea: mild (2-3 loose stools in 24 H), moderate (4-5 loose stools in 24 H), severe (>=6 in 24 H). For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by investigator or medically qualified person.
Time Frame: From Day 1 to Day 7 after vaccination
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo
Number analyzed (Participants) | 3678 | 3651
Percentage of participants
  Fever: >=38.0 degree C | 2.6 [2.1 to 3.1] | 2.9 [2.4 to 3.5]
  Fever: 38.0 to 38.4 degree C | 1.7 [1.3 to 2.1] | 1.5 [1.1 to 2.0]
  Fever: 38.5 to 38.9 degree C | 0.8 [0.5 to 1.1] | 1.2 [0.8 to 1.6]
  Fever: 39.0 to 40.0 degree C | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.3]
  Fever: >40.0 degree C | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.3]
  Fatigue: Any | 46.1 [44.5 to 47.7] | 43.8 [42.2 to 45.4]
  Fatigue: Mild | 23.5 [22.1 to 24.9] | 22.7 [21.4 to 24.1]
  Fatigue: Moderate | 21.3 [20.0 to 22.7] | 19.6 [18.4 to 21.0]
  Fatigue: Severe | 1.3 [1.0 to 1.8] | 1.4 [1.1 to 1.9]
  Fatigue: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Headache: Any | 31.0 [29.5 to 32.5] | 27.6 [26.2 to 29.1]
  Headache: Mild | 20.2 [18.9 to 21.5] | 17.9 [16.7 to 19.2]
  Headache: Moderate | 10.4 [9.4 to 11.4] | 9.4 [8.5 to 10.4]
  Headache: Severe | 0.4 [0.2 to 0.7] | 0.4 [0.2 to 0.6]
  Headache: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Nausea: Any | 20.0 [18.7 to 21.3] | 19.3 [18.0 to 20.6]
  Nausea: Mild | 14.4 [13.3 to 15.6] | 13.9 [12.8 to 15.0]
  Nausea: Moderate | 5.4 [4.7 to 6.1] | 5.2 [4.5 to 6.0]
  Nausea: Severe | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  Nausea: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Muscle pain: Any | 26.6 [25.1 to 28.0] | 17.1 [15.9 to 18.4]
  Muscle pain: Mild | 17.6 [16.4 to 18.9] | 10.0 [9.0 to 11.0]
  Muscle pain: Moderate | 8.6 [7.7 to 9.5] | 6.8 [6.0 to 7.7]
  Muscle pain: Severe | 0.4 [0.2 to 0.6] | 0.3 [0.2 to 0.6]
  Muscle pain: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Joint pain: Any | 11.6 [10.6 to 12.7] | 10.5 [9.5 to 11.6]
  Joint pain: Mild | 6.5 [5.7 to 7.3] | 6.0 [5.2 to 6.8]
  Joint pain: Moderate | 4.9 [4.2 to 5.7] | 4.4 [3.8 to 5.2]
  Joint pain: Severe | 0.2 [0.1 to 0.4] | 0.1 [0.0 to 0.2]
  Joint pain: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Vomiting: Any | 7.9 [7.0 to 8.8] | 7.0 [6.2 to 7.8]
  Vomiting: Mild | 6.4 [5.6 to 7.2] | 5.4 [4.7 to 6.1]
  Vomiting: Moderate | 1.3 [0.9 to 1.7] | 1.5 [1.2 to 2.0]
  Vomiting: Severe | 0.2 [0.1 to 0.4] | 0.1 [0.0 to 0.2]
  Vomiting: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]
  Diarrhea: Any | 11.3 [10.3 to 12.3] | 11.4 [10.4 to 12.5]
  Diarrhea: Mild | 9.1 [8.2 to 10.1] | 9.4 [8.4 to 10.4]
  Diarrhea: Moderate | 2.0 [1.6 to 2.5] | 1.9 [1.4 to 2.4]
  Diarrhea: Severe | 0.1 [0.0 to 0.3] | 0.2 [0.1 to 0.4]
  Diarrhea: Grade 4 | 0 [0.0 to 0.1] | 0 [0.0 to 0.1]

22. Primary Outcome: Percentage of Maternal Participants With AEs From the Time of Vaccination Through 1 Month After Vaccination (Safety)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were included in this outcome measure.
Time Frame: From vaccination on Day 1 up to 1 month after vaccination
Population: Maternal safety population included all randomized maternal participants who received investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo
Number analyzed (Participants) | 3698 | 3687
Percentage of participants | 14.0 [12.9 to 15.1] | 13.2 [12.2 to 14.4]

23. Primary Outcome: Percentage of Maternal Participants With SAEs Throughout the Study Period (Safety)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect or that was considered an important medical event.
Time Frame: From vaccination on Day 1 up to 6 months after delivery (maximum up to 10 months)
Population: Maternal safety population included all randomized maternal participants who received investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Maternal Participants: RSVpreF: Study-eligible pregnant women (maternal participants) were randomized to receive a single dose of 120 micrograms (mcg) RSVpreF, intramuscularly (IM) on Day 1 (day of vaccination). Participants were followed up to 6 months after delivery.
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo
Number analyzed (Participants) | 3698 | 3687
Percentage of participants | 16.6 [15.4 to 17.8] | 15.8 [14.6 to 17.0]

24. Secondary Outcome: Percentage of Infant Participants With Cases of Hospitalization Due to RSV Within 90, 120, 150, 180 and 360 Days After Birth (Efficacy)
Description: Results are reported as confirmed by endpoint adjudication committee.
Time Frame: Within 90, 120, 150, 180 and 360 days after birth
Population: as for outcome 2
Measure: Number; unit: %participants with hospitalization cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
%participants with hospitalization cases
  90 days after birth | 0.3 | 0.9
  120 days after birth | 0.4 | 1.1
  150 days after birth | 0.5 | 1.2
  180 days after birth | 0.6 | 1.3
  360 days after birth | 1.4 | 1.9
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 90 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 69.7, 95% CI 2-sided [37.1 to 86.7]
Statistical Analysis 2: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 120 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 61.5, 95% CI 2-sided [28.6 to 80.3]
Statistical Analysis 3: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 150 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 57.1, 95% CI 2-sided [23.9 to 76.8]
Statistical Analysis 4: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 180 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 55.3, 95% CI 2-sided [23.8 to 74.6]
Statistical Analysis 5: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 360 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 24.2, 95% CI 2-sided [-11.1 to 48.6]

25. Secondary Outcome: Percentage of Infant Participants With MA-LRTI Cases Due to Any Cause With Protocol Defined Criteria Occurring Within 90, 120, 150, 180 and 360 Days After Birth (Efficacy)
Description: MA-LRTI cases due to any cause was defined as an infant with a MA-RTI visit with age related fast breathing (RR >=60 bpm for <2 months of age [<60 days of age], >=50 bpm for >=2 months to <12 months of age, or >=40 bpm for >=12 months to 24 months of age) or SpO2 <95% or chest wall indrawing.
Time Frame: Within 90, 120, 150, 180 and 360 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases
  90 days after birth | 5.6 | 6.2
  120 days after birth | 8.1 | 8.8
  150 days after birth | 10.3 | 11.3
  180 days after birth | 12.4 | 13.0
  360 days after birth | 17.5 | 18.4
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 90 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 9.5, 95% CI 2-sided [-10.1 to 25.7]
Statistical Analysis 2: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 120 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 6.7, 95% CI 2-sided [-9.8 to 20.7]
Statistical Analysis 3: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 150 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 7.7, 95% CI 2-sided [-6.5 to 20.1]
Statistical Analysis 4: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 180 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 4.1, 95% CI 2-sided [-9.5 to 16.0]
Statistical Analysis 5: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy within 360 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 4.6, 95% CI 2-sided [-6.6 to 14.6]

26. Secondary Outcome: Percentage of Infant Participants With MA-LRTI Cases Due to RSV Occurring Within 210, 240, 270 and 360 Days After Birth (Efficacy)
Description: as for outcome 2
Time Frame: Within 210, 240, 270 and 360 days after birth
Population: as for outcome 2
Measure: Number; unit: % of participants with MA-LRTI cases
Arm/Group | Infant Participants: RSVpreF | Infant Participants: Placebo
Number analyzed (Participants) | 3585 | 3563
% of participants with MA-LRTI cases
  210 days after birth | 2.3 | 4.0
  240 days after birth | 2.5 | 4.2
  270 days after birth | 2.8 | 4.4
  360 days after birth | 3.4 | 5.1
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy at 210 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 43.8, 95% CI 2-sided [25.6 to 57.7]
Statistical Analysis 2: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy at 240 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 39.7, 95% CI 2-sided [21.3 to 54.1]
Statistical Analysis 3: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy at 270 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 35.0, 95% CI 2-sided [16.1 to 49.9]
Statistical Analysis 4: Comparison: Infant Participants: RSVpreF vs Infant Participants: Placebo; Vaccine efficacy at 360 days after birth. Vaccine efficacy was calculated as 1-(P/[1-P]), where P is the number of cases in the RSVpreF group divided by the total number of cases. The confidence interval was adjusted using Bonferroni procedure and accounting for the primary endpoints results. Vaccine efficacy was presented in percentage; Test type: Other; Vaccine efficacy = 33.0, 95% CI 2-sided [15.2 to 47.1]

ADVERSE EVENTS:
Time Frame: Maternal participants: Local reactions and systemic events: From Day 1 to Day 7 after vaccination; SAEs: From vaccination on Day 1 up to 6 months after delivery (maximum up to 10 months); Non-SAEs: From vaccination on Day 1 up to 1 month after vaccination; Infant participants: SAEs: From birth up to 24 months of age; Non-SAEs: From birth up to 1 month after birth
Description: Local reactions and Systemic events were assessed by systematic assessment and non-SAEs and SAE by non-systematic events. Same event may appear as both an SAE and non-SAE. But what is presented are distinct events. An event may be categorized as serious in one participant & as non-serious in another, or a participant may have experienced both SAE & non-SAE. Maternal & infant safety population was evaluated.
Arm/Group | Maternal Participants: RSVpreF | Maternal Participants: Placebo | Infant Participants: RSVpreF | Infant Participants: Placebo
All-Cause Mortality (participants affected / at risk) | 1/3698 | 0/3687 | 8/3659 | 14/3646
Serious Adverse Events (participants affected / at risk) | 613/3698 | 581/3687 | 697/3659 | 689/3646
Other Adverse Events (participants affected / at risk) | 2755/3698 | 2339/3687 | 674/3659 | 598/3646
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Participants: RSVpreF (N=3698) | Maternal Participants: Placebo (N=3687) | Infant Participants: RSVpreF (N=3659) | Infant Participants: Placebo (N=3646)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 2
Device occlusion (Product Issues) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 3 | 23 | 18
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 6 | 3
Inborn error of metabolism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 29 | 31
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | 7
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8 | 7
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 29 | 33 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 49 | 42
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Sepsis neonatal (Infections and infestations) | 0 | 0 | 19 | 21
Skull base tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 3
Ventricular hypoplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Amniotic fluid volume decreased (Investigations) | 2 | 0 | 0 | 0
Apgar score low (Investigations) | 0 | 0 | 0 | 1
Base excess decreased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Blood glucose (Investigations) | 0 | 0 | 1 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0
Body temperature fluctuation (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 4 | 2
Cardiovascular function test abnormal (Investigations) | 0 | 0 | 1 | 0
Cholangiogram abnormal (Investigations) | 0 | 1 | 0 | 0
Cytomegalovirus test positive (Investigations) | 0 | 1 | 0 | 0
Foetal heart rate abnormal (Investigations) | 7 | 2 | 0 | 0
Foetal heart rate indeterminate (Investigations) | 1 | 1 | 0 | 0
Foetal monitoring abnormal (Investigations) | 3 | 6 | 0 | 0
HIV test positive (Investigations) | 1 | 0 | 1 | 0
Nutritional condition abnormal (Investigations) | 0 | 0 | 3 | 0
Oxygen saturation abnormal (Investigations) | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 3 | 3
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 5 | 2 | 0 | 3
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 1
Ultrasound antenatal screen abnormal (Investigations) | 1 | 2 | 0 | 0
Ultrasound foetal abnormal (Investigations) | 0 | 3 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 3 | 1
Bradycardia foetal (Cardiac disorders) | 8 | 13 | 0 | 0
Bradycardia neonatal (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac ventricular disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 1 | 0 | 0
Foetal arrhythmia (Cardiac disorders) | 2 | 0 | 0 | 0
Foetal heart rate deceleration abnormality (Cardiac disorders) | 6 | 12 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1
Neonatal bradyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 37 | 30 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 3 | 5
Pulmonary valve thickening (Cardiac disorders) | 0 | 0 | 1 | 0
Right atrial enlargement (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 4 | 2 | 0 | 1
Tachycardia foetal (Cardiac disorders) | 2 | 3 | 0 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 3
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Aberrant aortic arch (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Accessory spleen (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Anal atresia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Anisomelia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Anomaly of external ear congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Anorchism (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Anorectal malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 37 | 46
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Autosomal chromosome anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 0
Bifid ureter (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Brachycephaly (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 1
Branchial cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Cataract congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Chordee (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 3
Chromosomal deletion (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Cleft lip and palate (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Cleft palate (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Cleft uvula (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 2
Coloboma (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Congenital aortic anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital cytomegalovirus infection (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Congenital diaphragmatic eventration (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital eye disorder (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 3
Congenital hypothyroidism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 2
Congenital knee deformity (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital megacolon (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital melanocytic naevus (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Congenital musculoskeletal disorder (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital musculoskeletal disorder of spine (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital pulmonary artery anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital retinoblastoma (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 5
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 1
Congenital torticollis (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Congenital urethral anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Craniofacial deformity (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 12 | 18
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Deafness congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 11 | 15
Dextrocardia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Dolichocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Duane's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Ear malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Eyelid ptosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 3
Galactosaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Gallbladder anomaly congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Genitalia external ambiguous (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Hypoplastic left heart syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 6 | 11
Intestinal malrotation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Iris coloboma (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Kidney duplex (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Laryngeal cleft (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 1
Left-to-right cardiac shunt (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Limb reduction defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Macrocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 5 | 3
Meningocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Microcephaly (Congenital, familial and genetic disorders) | 0 | 0 | 7 | 7
Micrognathia (Congenital, familial and genetic disorders) | 0 | 0 | 5 | 2
Micropenis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Microphthalmos (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Mitochondrial encephalomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Naevus flammeus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Neurofibromatosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3
Oesophageal atresia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Optic nerve hypoplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Osteochondrodysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 13 | 14
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Penile torsion (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 3
Penoscrotal fusion (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 4
Phenylketonuria (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3
Poland's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Polycystic liver disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 7
Posterior segment of eye anomaly congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Preternatural anus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 7 | 6
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 1
Pyruvate carboxylase deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Renal aplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 2
Renal dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Reproductive tract hypoplasia, male (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Scaphocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Septo-optic dysplasia (Congenital, familial and genetic disorders) | 0 | 0 (0) | 1 | 0
Spina bifida occulta (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Supernumerary nipple (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Syndactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 5 | 4
Tethered oral tissue (Congenital, familial and genetic disorders) | 0 | 0 | 18 | 16
Thalassaemia alpha (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 2
Vallecular cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Vascular malformation (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 15 | 21
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 1 | 4
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemolysis neonatal (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Idiopathic neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Polycythaemia neonatorum (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Splenic cyst (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Atypical migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Benign enlargement of the subarachnoid spaces (Nervous system disorders) | 0 | 0 | 3 | 2
Cerebral cyst (Nervous system disorders) | 0 | 0 | 3 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 5 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalomalacia (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy neonatal (Nervous system disorders) | 0 | 0 | 2 | 3
Epilepsy (Nervous system disorders) | 0 | 1 | 2 | 0
External hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 9 | 13
Headache (Nervous system disorders) | 2 | 2 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 1
Intracranial haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 1 | 2
Lenticulostriatal vasculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Motor developmental delay (Nervous system disorders) | 0 | 0 | 2 | 0
Moyamoya disease (Nervous system disorders) | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 2 | 2
Neurodevelopmental delay (Nervous system disorders) | 0 | 0 | 0 | 1
Non-epileptic paroxysmal event (Nervous system disorders) | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 3 | 6
Speech disorder developmental (Nervous system disorders) | 0 | 0 | 2 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0
Subdural haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 0 | 1
Subependymal cyst (Nervous system disorders) | 0 | 0 | 3 | 3
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Tethered cord syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 2 | 1
Pupillary disorder (Eye disorders) | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Brief resolved unexplained event (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 3
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 10 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal flaring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Neonatal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 11 | 14
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 11 | 14
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 49 | 46
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 8
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 33 | 29
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Food protein-induced enterocolitis syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 5
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 3
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 6 | 8
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Meconium ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Meconium plug syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Terminal ileitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 5
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 6 | 9
Hydroureter (Renal and urinary disorders) | 0 | 0 | 0 | 1
Kidney small (Renal and urinary disorders) | 0 | 0 | 1 | 1
Neonatal anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrectasia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 6 | 8
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureterocele (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 2 | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Ankle deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Head deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint noise (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Retrognathia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 7
Hypopituitarism (Endocrine disorders) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 9 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 6 | 5
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Food aversion (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 20 | 17
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 13 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 1
Abscess oral (Infections and infestations) | 0 | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Amniotic cavity infection (Infections and infestations) | 10 | 5 | 0 | 0
Amoebic dysentery (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 2 | 2
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 3 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0
Botulism (Infections and infestations) | 0 | 0 | 1 | 0
Breast abscess (Infections and infestations) | 1 | 4 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 4
Cellulitis (Infections and infestations) | 1 | 0 | 3 | 2
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Chest wall abscess (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Endometritis (Infections and infestations) | 5 | 2 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 14 | 15
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Mastitis (Infections and infestations) | 5 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 2
Meningitis cronobacter (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis enteroviral (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Neonatal infection (Infections and infestations) | 0 | 0 | 1 | 3
Neonatal infective mastitis (Infections and infestations) | 0 | 0 | 0 | 1
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 3 | 1
Omphalitis (Infections and infestations) | 0 | 0 | 4 | 2
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 2
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 3 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 0
Pathogen resistance (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pilonidal disease (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 2 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 5 | 0 | 0
Postpartum sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Puerperal infection (Infections and infestations) | 1 | 3 | 0 | 0
Puerperal pyrexia (Infections and infestations) | 1 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 4 | 2 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 3 | 1
Pyomyositis (Infections and infestations) | 0 | 0 | 0 | 1
Pyuria (Infections and infestations) | 0 | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 1
Secondary syphilis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 9 | 4
Septic coagulopathy (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 0 | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 6 | 15 | 14
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bladder injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Electrical burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Fractured skull depressed (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury to brachial plexus due to birth trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Maternal drugs affecting foetus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Perineal injury (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 4
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Eye haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Eyelid haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 5
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Juvenile xanthogranuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Spinal cord lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ulcerated haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Extradural haematoma evacuation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 0 | 1 | 0 | 0
Cyanosis (Vascular disorders) | 0 | 0 | 0 | 5
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 13 | 6 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 1
Kawasaki's disease (Vascular disorders) | 0 | 0 | 1 | 1
Scalp haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 0 | 2
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 2 | 1
Drug withdrawal syndrome neonatal (General disorders) | 0 | 0 | 3 | 0
Fever neonatal (General disorders) | 0 | 0 | 2 | 1
Hypertrophy (General disorders) | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 4 | 2
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Macrosomia (General disorders) | 0 | 1 | 0 | 2
Mass (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 2 | 8
Abnormal labour (Pregnancy, puerperium and perinatal conditions) | 5 | 7 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 37 | 43 | 0 | 0
Birth trauma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 6 | 5 | 0 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 14 | 19 | 0 | 0
Delayed delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 7 | 3 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Face presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 4 | 0 | 0
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 9 | 8 | 0 | 0
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 1 | 5 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 6 | 8 | 0 | 0
Foetal disorder (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 67 | 65 | 1 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 15 | 11 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 5 | 4 | 0 | 0
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 6 | 7 | 0 | 0
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 0 | 0
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Foetal vascular malperfusion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Foetal-maternal haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 43 | 41 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 2 | 3 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 7 | 3 | 0 | 0
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Hypoxic ischaemic encephalopathy neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 3 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 77 | 69
Labour complication (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 2
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 0 | 0
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 5 | 5 | 0 | 1
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 15 | 12 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 16 | 21 | 0 | 0
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Placental calcification (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 2 | 4 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 67 | 53 | 0 | 0
Precipitate labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 30 | 24 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 15 | 9 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 14 | 16 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 19 | 13 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 15 | 11 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 23 | 21 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 9 | 7 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 10 | 10 | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 8 | 5 | 0 | 0
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 0 | 0
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 6 | 10
Spontaneous rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 4 | 1 | 0 | 0
Superimposed pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 15 | 14 | 0 | 0
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 3 | 3
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 0 | 0
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 5 | 3 | 0 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 3 | 0 | 0
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Uterine tachysystole (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Disease risk factor (Social circumstances) | 0 | 0 | 0 | 1
ABO incompatibility (Immune system disorders) | 0 | 0 | 1 | 4
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 2
Blood type incompatibility (Immune system disorders) | 0 | 0 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 0
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 1
Rhesus incompatibility (Immune system disorders) | 1 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 4 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 3 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 2 | 1 | 0
Cholestasis of pregnancy (Hepatobiliary disorders) | 11 | 6 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 51 | 42
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Intrahepatic portal hepatic venous fistula (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Neonatal cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Perineal disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular retraction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Threatened uterine rupture (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Uterine cervix hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine disorder (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Vulval haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Brief psychotic disorder, with postpartum onset (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0
Panic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Perinatal depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Selective eating disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Maternal Participants: RSVpreF (N=3698) | Maternal Participants: Placebo (N=3687) | Infant Participants: RSVpreF (N=3659) | Infant Participants: Placebo (N=3646)
SARS-CoV-2 test positive (Investigations) | 148 | 114 | 119 | 108
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 49 | 30
Tethered oral tissue (Congenital, familial and genetic disorders) | 0 | 0 | 41 | 32
Headache (HEADACHE) (Nervous system disorders) | 1141/3678 | 1009/3651 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 414/3678 | 416/3651 | 0/3569 | 0
Nausea (NAUSEA) (Gastrointestinal disorders) | 734/3678 | 705/3651 | 0 | 0
Vomiting (VOMITING) (Gastrointestinal disorders) | 289/3678 | 254/3651 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 31 | 39
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 265/3678 | 8/3651 | 0 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 426/3678 | 384/3651 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 977/3678 | 626/3651 | 0 | 0
Fatigue (FATIGUE) (General disorders) | 1696/3678 | 1599/3651 | 0 | 0
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 1496/3678 | 371/3651 | 0 | 0
Pyrexia (FEVER) (General disorders) | 94/3678 | 107/3651 | 0 | 0
Swelling (SWELLING) (General disorders) | 228/3678 | 8/3651 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 191 | 183
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 157 | 127
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 158 | 130
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 182 | 153 | 0 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 59 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04424316/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT04424316/SAP_001.pdf